CLINICAL TRIAL: NCT06030583
Title: An Investigation of Vocal Hygiene, Vocal Behaviors, and Quality of Life Associated With Voice in Children With and Without Attention Deficit Hyperactivity Disorder
Brief Title: The Investigation of Vocal Behaviors in Children With ADHD
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özlem Beşik Topçu, Principal Investigator, Hacettepe University
Other Study IDs: HUSLP_ADHD_VOICE
Record Dates: First submitted 2023-08-30; First posted 2023-09-11 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-01

CONDITIONS: Voice Disorders in Children; Voice
Keywords: voice disorders in children; ADHD; attention deficit and hyperactivity disorder; vocal behaviors in children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: The research group comprises children aged 8 to 11 diagnosed with Attention Deficit Hyperactivity Disorder.
  Interventions: Other: Scales and Forms
- Control Group: The control group consists of children aged 8 to 11 who do not have a diagnosis of ADHD, matched in terms of age and gender with the research group.
  Interventions: Other: Scales and Forms

INTERVENTIONS:
Other: Scales and Forms — This study does not involve any interventions. Information will be collected from the study group and the control group through scales and forms.

SUMMARY:
The aim is to gain information about vocal hygiene knowledge level, phonotrauma behavior frequency, voice-related quality of life, and voice handicap index scores in children diagnosed with ADHD aged 8 to 11, through inter-group comparisons of scale and questionnaire data between children diagnosed with ADHD and control group participants aged 8 to 11.

DETAILED DESCRIPTION:
The study will include children aged 8 to 11 with and without a diagnosis of Attention Deficit Hyperactivity Disorder (ADHD). The study and control groups have been determined with age and gender matching.

Within the scope of the study, a comparison between groups will be conducted through the scores of the Vocal Hygiene Awareness form, Pediatric Phonotrauma Assessment Questions for Parents, Voice Related Quality of Life Survey, and the Teacher-Reported Pediatric Voice Handicap Index to examine whether there are any differences between the groups. The Vocal Hygiene Awareness form will be completed by the child. The Pediatric Phonotrauma Assessment Questions for Parents, Voice Related Quality of Life Survey, and the Pediatric Voice Handicap Index will be completed by the parents. The Teacher-Reported Pediatric Voice Handicap Index will be filled out by the child's teacher.

The number of participants to be included in the study has been calculated using G Power 3.1 program. Based on an analysis with a power of 0.80 and α (type 1 error) = 0.05 using an independent t-test, 42 participants for each group, totaling 84 participants, are planned to be included in the study. Data analysis will be carried out using IBM SPSS Statistics 23 program. Firstly, the normal distribution of ordinal variables will be tested. If the assumption of normality is met, parametric tests will be used; otherwise, non-parametric tests will be employed. A statistical significance value of p < 0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* For study group

  * Having been diagnosed with ADHD according to DSM-5 (The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) diagnostic criteria
  * Being in the age range of 8-11
  * Having Turkish as the native language
  * To have a score below the cut-off score (<13) on the Turkish Pediatric Voice Handicap Index.

For the control group:

* Not having any psychiatric diagnosis
* Being in the age range of 8-11
* Having Turkish as the native language
* To have a score below the cut-off score (<13) on the Turkish Pediatric Voice Handicap Index.

Exclusion Criteria:

* For the research group;

  * Having any history of upper respiratory tract infection in the period up to two weeks before the data collection date (one of the questionnaire requests considering the last two-week period as a reference).
  * Having any known neurological, systemic, or endocrinological diseases affecting the voice.
  * Having undergone vocal surgery or received voice therapy.
  * Having a diagnosis of current hearing loss.
  * Having comorbid autism spectrum disorder, intellectual disability, language, and speech disorders.
  * The family or the child not wanting to participate in the study.

For the control group;

* Having any history of upper respiratory tract infection in the period up to two weeks before the data collection date.
* Having any known neurological, systemic, or endocrinological diseases affecting the voice.
* Having undergone vocal surgery or received voice therapy.
* Having a diagnosis of current hearing loss.
* Having a neurological or psychiatric diagnosis.
* Having a diagnosis of language and speech disorders.
* The family or the child not wanting to participate in the study.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study group participants will be comprised of children aged 8 to 11 who have been diagnosed with ADHD in the Department of Child and Adolescent Psychiatry at Hacettepe University. Their inclusion in the study will be based on voluntary participation. For the control group, participants will be reached through the snowball sampling method, with age and gender matching, and their inclusion in the study will also be based on voluntary participation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Inter-group Differences Associated with Phonotraumatic Behaviors | The process of collecting data from participants once takes approximately 30 minutes
  Scores Obtained from Pediatric Phonotrauma Assessment Questions for Parents
Inter-group Differences Associated with Vocal Hygiene Knowledge | The process of collecting data from participants once takes approximately 30 minutes
  Scores Obtained from Questions on Vocal Hygiene Awareness

SECONDARY OUTCOMES:
Inter-group Differences Associated with Voice Related Quality of Life Survey | The process of collecting data from participants once takes approximately 30 minutes
  Scores Obtained from the Voice Related Quality of Life Survey
Inter-group Differences Associated with the Teacher-Reported Pediatric Voice Handicap Index | The process of collecting data from participants once takes approximately 30 minutes
  Scores Obtained from the Teacher-Reported Pediatric Voice Handicap Index

CONTACTS AND LOCATIONS:
Overall Officials: Esra Özcebe, Professor, Study Director — Istanbul University- Cerrahpaşa, Audiology Department; Fatma Esen Aydınlı, Assoc. Prof., Study Chair — Hacettepe University, Speech and Language Therapy Departmant; Özlem Beşik Topçu, SLP, Study Chair — Hacettepe University, Speech and Language Therapy; Meltem Çiğdem Kirazlı, Ph.D., Study Chair — Hacettepe University, Speech and Language Therapy; Nur Seda Saban Dülger, SLP, Study Chair — Hacettepe University, Speech and Language Therapy; Merve Öğülmüş Uysal, SLP, Study Chair — Hacettepe University, Speech and Language Therapy; Halime Tuna Çak Esen, Assos. Prof., Study Chair — Independent Researcher; Cihan Aslan, Dr., Study Chair — Hacettepe University Faculty of Medicine Department of Pediatric Mental Health And Diseases
Locations (1):
- Hacettepe University, Speech and Language Therapy, Ankara, Turkey (Türkiye)